CLINICAL TRIAL: NCT00974168
Title: A Phase II Trial Evaluating the Efficacy of a Radio-Biological Based Re-Irradiation Strategy for Patients With Malignant Spinal Cord Compression
Brief Title: Spinal Cord Compression Re-Treat Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 07-11; ICORG 07-11; EU-20953; NCT00624507 (obsolete NCT alias)
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2018-07

CONDITIONS: Pain; Radiation Toxicity; Spinal Cord Compression; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: pain; radiation toxicity; spinal cord compression; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Pain; Radiation Injuries; Spinal Cord Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Radiation Cumulative BED ≤ 100 Gy2
  Interventions: Radiation: Cumulative BED ≤ 100
- B (Active Comparator): Cumulative BED ≤ 130 Gy2
  Interventions: Radiation: Cumulative BED ≤ 130 Gy2

INTERVENTIONS:
Radiation: Cumulative BED ≤ 100 — Radiation
  Arms: A
Radiation: Cumulative BED ≤ 130 Gy2 — Radiation
  Arms: B

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Radiation therapy may be effective in treating malignant spinal cord compression in patients who have received previous radiation therapy to the spine.

PURPOSE: This phase II trial is studying radiation therapy in treating patients with malignant spinal cord compression.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of a biologically effective dose-based re-irradiation strategy, in terms of the response rate (based on the mobility score using the Tomita scale where improvement in mobility or stable mobility score will be regarded as a response) in patients with malignant spinal cord compression.

Secondary

* To determine quality of life as assessed by the EORTC QLQ-C15 PAL version 1.0 questionnaire.
* To determine the non-spinal radiation-induced toxicity using standard RTOG criteria.
* To determine the rate of long-term spinal toxicity and radiation-induced myelopathy using the RTOG SOMA morbidity grading system.

OUTLINE: Patients are divided into 2 groups according to the interval since their most recent radiotherapy to the involved area of the spinal cord.

* Group 1 (< 6 months since prior radiotherapy): Patients undergo radiotherapy for a cumulative biologically effective dose (BED) ≤ 100 Gy_2 in addition to receiving other current treatment.
* Group 2 (≥ 6 months since prior radiotherapy): Patients undergo radiotherapy for a cumulative BED ≤ 130 Gy_2 in addition to receiving other current treatment.

Mobility score is assessed and patients complete a quality-of-life assessment at baseline and at each follow-up visit starting at week 5.

After completion of study treatment, patients are followed up at 1 and 5 weeks, at 3 months, and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* MRI-confirmed diagnosis of malignant spinal cord compression

  * MRI of the entire spine performed
* Histologically proven malignancy

  * No primary tumors of the spine or vertebral column
* Undergone previous radiotherapy to the involved area of the spinal cord (e.g., full segment and/or ≥ 2 cm in cranio-caudal of overlap between the 2 areas treated)

  * Maximum biologically effective dose received from previous irradiation ≤ 90 Gy_2
* Deemed not suitable for neurosurgical intervention at the time of initial assessment

  * Patients deemed inoperable are eligible

PATIENT CHARACTERISTICS:

* Karnofsky performance status 40-100%
* Short life expectancy
* No medical or psychiatric condition that, in the opinion of the investigator or research team, contraindicates participation in this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-10; Primary Completion 2016-12 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Response to treatment as assessed by mobility via the Tomita mobility scale | 5 weeks after completion of radiation therapy
Overall response rate (stabilization and response) (stage I) | 5 weeks subsequent to radiation therapy and 3 monthly timepoints thereafter

SECONDARY OUTCOMES:
Incidence of radiation-induced myelopathy via the RTOG SOMA morbidity grading system | 5 weeks subsequent to radiation therapy and 3 monthly timepoints thereafter
Toxicity other than spine (acute toxicity assessed at weeks 1 and 5 and late toxicity assessed at 3 months and at subsequent follow-ups) evaluated according to RTOG criteria | 5 weeks subsequent to radiation therapy and 3 monthly timepoints thereafter
Pain control via the pain visual analogue score | 5 weeks subsequent to radiation therapy and 3 monthly timepoints thereafter
Quality of life via the EORTC QLQ-C15 PAL version 1.0 questionnaire | 5 weeks subsequent to radiation therapy and 3 monthly timepoints thereafter
Median survival (time from the date of recruitment/treatment to death) | Until death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Thirion, Dr, Principal Investigator — Saint Luke's Hospital
Locations (2):
- Ireland (2):
  - Saint Luke's Radiation Oncology Network, Dublin
  - Galway University Hospital, Galway

REFERENCES:
- [Derived] Wallace ND, Dunne MT, McArdle O, Small C, Parker I, Shannon AM, Clayton-Lea A, Parker M, Collins CD, Armstrong JG, Gillham C, Coffey J, Fitzpatrick D, Salib O, Moriarty M, Stevenson MR, Alvarez-Iglesias A, McCague M, Thirion PG. Efficacy and toxicity of primary re-irradiation for malignant spinal cord compression based on radiobiological modelling: a phase II clinical trial. Br J Cancer. 2023 Feb;128(4):576-585. doi: 10.1038/s41416-022-02078-w. Epub 2022 Dec 8. PMID 36482188